CLINICAL TRIAL: NCT02911051
Title: Clinical Study Evaluating the Safety of a New Catheter for Urinary Intermittent Catheterization in Self Catheterized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OPM-G-H-1303; 2014-A01774-43-A (Other: French Health Autority)
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Intermittent Urethral Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Actreen Hydrolite Cath (Experimental): a new hydrophilic coated catheter for Urinary Intermittent Catheterisation
  Interventions: Device: Actreen Hydrolite Cath

INTERVENTIONS:
Device: Actreen Hydrolite Cath — Depending of the use of the self catheterized patient could be 4 to 6 Actreen Hydrolite Cath per day

SUMMARY:
The clinical study evaluates the safety of a new catheter for Urinary Intermittent Catheterisation in self catheterized patients

ELIGIBILITY:
Inclusion Criteria:

1. male patient
2. patient is at least 18 years old
3. patient having normal or impaired sensation in the urethra
4. patient catheterizing at least 4 times a day
5. patient using Ch 12 or 14 catheter for self clean urinary catheterization
6. patient using a Nelaton catheter for self clean urinary catheterization
7. patient using self clean urinary catheterization for at least one month
8. patient covered with social insurance

Exclusion Criteria:

1. patient having a symptomatic urinary tract infection as assessed by the investigator (5 days after end of treatment for UTI, patient can be considered by the investigator for inclusion)
2. patient with urethral hypersensitivity
3. patient being mentally unstable not being assessed by the investigator as capable to follow the study procedure
4. patient already participating in another clinical study or who have previously participated in this investigation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Safety of Hydrolite Cath will be demonstrated by listing any adverse event(s) related to the use of Actreen® Hydrolite Cath and other occurrence | All adverse event(s) occured during the 7 (±1) days, related to the use of Actreen Hydrolite Cath, will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Chartier-Kastler Emmanuel, Principal Investigator — Hôspital Raymond Poincaré - Garches
Locations (1):
- Chartier-Kastler, Garches, France

IPD SHARING:
Plan to Share IPD: No